CLINICAL TRIAL: NCT04763824
Title: KanSurvive: Testing a Model for Improving Cancer Survivorship Care in Rural Practice
Acronym: KANSURVIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Klemp, PhD, MA, MPH, Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00144314; 5R01CA240103-02 (NIH)
Record Dates: First submitted 2020-11-25; First posted 2021-02-21 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer
Keywords: Cancer Survivorship; Rural Primary Care Practices
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility study aimed at evaluating the effectiveness of the KanSurvive ECHO intervention combined with practice facilitation to promote the adoption of evidence-based practice survivorship care guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KanSurvive Telementoring with Practice Facilitation (Other): This study does not involve a therapeutic intervention.
  The KanSurvive project includes Project ECHO telementoring and education with practice facilitation to improve the delivery of cancer survivorship care in primary care practice.
  Interventions: Other: KanSurvive ECHO and Practice Facilitation

INTERVENTIONS:
Other: KanSurvive ECHO and Practice Facilitation — Four, 1-hour, virtual, case-based education sessions covering the evidence-based practice guidelines for breast, colorectal, lung, and prostate cancer survivorship care. Practice facilitation also provided to support participating primary care practices with quality improvement in the delivery of cancer survivorship care.

SUMMARY:
Approximately, 20 rural primary care practices to participate in a delayed intervention-controlled trial.

Phase I: Formal and structured work flow evaluations to better identify specific gaps in processes of care while assessing what on-going training is needed for adoption of high-quality cancer survivorship care in rural practice. These will be incorporated into the ECHO sessions (Aim 1).

Phase II: Conduct and test the effectiveness of the novel KanSurvive-ECHO intervention (Aim 2) and finally identify barriers and facilitators to implementation of KanSurvive-ECHO (Aim 3).

DETAILED DESCRIPTION:
While evidence-based practice (EBP) guidelines exist for cancer survivorship care, implementation in rural practices has fallen short. Approximately 72.5% of Kansas cancer survivors who have completed their cancer treatment receive a majority of their health care from Primary Care Providers, yet these providers describe a lack of basic awareness of risk-based surveillance, effects of cancer treatment and their management, as well as inadequate resources, and growing administrative demands as reasons for not working to improve survivorship care. These factors may also prevent shared care management of cancer survivors between primary care and rural oncology care providers. There is a pressing need to understand primary care practice capacity to implement guideline informed management and follow-up for cancer survivors in the acute and extended phases of care.

Specific Aim 1. Formally assess gaps in processes of care and additional training needed to result in actual adoption of high-quality care for acute and chronic survivors of breast, colorectal, lung, and prostate cancer in 20 rural primary care practices. Utilize this formative information to further refine the KanSurvive-ECHO.

Specific Aim 2. Evaluate the effectiveness of KanSurvive-ECHO for enhancing evidence-based survivorship care for rural breast, colorectal, lung, and prostate cancer survivors.

Hypothesis: Compared to delayed intervention control, rural primary care practices randomized to KanSurvive-ECHO will demonstrate greater concordance with evidence-based survivorship care guidelines as measured by a composition score determined by change in EHR documentation consistent with guideline concordant care.

Specific Aim 3: Utilizing the Integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework describe key facilitators and barriers to implementation of KanSurvive-ECHO including innovation, recipients, context, and facilitation.

This novel project will provide a model for development of a community of practice using practice facilitation and Project ECHO to improve the management and follow-up of cancer survivors in the acute and extended phases of cancer survivorship.

ELIGIBILITY:
Inclusion Criteria:

1. Primary care practice (PCP) caring for rural cancer survivors
2. Willing to participate in four ECHO sessions
3. Capable and willing to complete pre- and post- data collection under a data use agreement
4. Cancer survivor data is eligible for extraction if the patient is a breast, prostate, lung, and/or colorectal cancer survivor and considered to have a "reasonable likelihood" of 24-month survival by a practice provider.

Exclusion Criteria:

1. PCPs unwilling to engage in project activities
2. PCPs with no rural-dwelling patients on their patient panel
3. Cancer survivor data is ineligible for extraction if the patient is <18 years of age or >75 years of age, is currently receiving hospice services, or has a history of cancer other than breast, prostate, lung, or colorectal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Cancer Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinics were the unit of assignment. The intervention was delivered at the clinic level. Outcome data were collected through retrospective, de-identified EHR chart reviews. Participants represent chart abstractions for cancer survivors seen during two independent audit periods: a baseline (pre-intervention) chart audit and a 24-month post-intervention chart audit. These audit samples were drawn from the same participating clinics but do not represent the same individual cancer survivors.
Groups:
- Baseline (Pre-Intervention) Chart Audit: This arm represents the baseline, pre-intervention chart audit sample drawn from participating primary care clinics. Charts included in this audit reflect an independent analytic sample of cancer survivors being seen in the practice. Demographic characteristics were abstracted at this time point to describe the baseline sample. Analyses are descriptive and no inferential comparisons were conducted between baseline and post-intervention samples.
- 24-Month (Post-Intervention) Follow-Up Chart Audit: This arm represents the analytic sample of EHR charts reviewed at the 24-month post-intervention time point. Charts reflect an independent sample drawn from the same participating clinics and do not necessarily represent the same cancer survivors included in the baseline chart audit.
Period: Baseline Arm
Arm/Group | Baseline (Pre-Intervention) Chart Audit | 24-Month (Post-Intervention) Follow-Up Chart Audit
Started (Follow-Up EHR Chart Review Data) | 138 (Participants represent independent EHR chart audit samples drawn from the same participating clinics at different time points. Individuals included in the baseline (pre-intervention) chart audit are not necessarily the same cancer survivors included in the 24-month post-intervention chart audit. Therefore, the number of participants starting the post-intervention period is not expected to equal the number who completed the baseline period.) | 0 (Participants represent independent EHR chart audit samples drawn from the same participating clinics at different time points. Individuals included in the baseline (pre-intervention) chart audit are not necessarily the same cancer survivors included in the 24-month post-intervention chart audit. Therefore, the number of participants starting the post-intervention period is not expected to equal the number who completed the baseline period.)
Completed | 138 | 0
Not Completed | 0 | 0
Period: Post-Intervention Arm
Arm/Group | Baseline (Pre-Intervention) Chart Audit | 24-Month (Post-Intervention) Follow-Up Chart Audit
Started | 0 (Participants represent independent EHR chart audit samples drawn from the same participating clinics at different time points. Individuals included in the baseline (pre-intervention) chart audit are not necessarily the same cancer survivors included in the 24-month post-intervention chart audit. Therefore, the number of participants starting the post-intervention period is not expected to equal the number who completed the baseline period.) | 129 (Participants represent independent EHR chart audit samples drawn from the same participating clinics at different time points. Individuals included in the baseline (pre-intervention) chart audit are not necessarily the same cancer survivors included in the 24-month post-intervention chart audit. Therefore, the number of participants starting the post-intervention period is not expected to equal the number who completed the baseline period.)
Completed | 0 | 129
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: "Participants" represent EHR charts selected for analysis from participating primary care clinics. Charts were abstracted during two independent audit periods-baseline (pre-intervention) and 24-month post-intervention-and do not represent the same individual cancer survivors followed longitudinally. No human participants were prospectively enrolled.
Groups:
- Baseline (Pre-Intervention) Chart Audit: This arm represents the baseline, pre-intervention chart audit sample drawn from participating primary care clinics prior to implementation of the KanSurvive ECHO + Practice Facilitation intervention.
  Charts included in this audit reflect an independent analytic sample of cancer survivors and do not necessarily represent the same individuals included in the baseline chart audit.
  Demographic characteristics were abstracted at this time point (Baseline) to describe the post-intervention sample.
  Analyses are descriptive and no inferential comparisons were conducted between baseline and post-intervention samples.
- 24-Month Follow-Up (Post-Intervention) Chart Audit: This arm represents the 24-month post-intervention chart audit sample drawn from the same participating primary care clinics following implementation of the KanSurvive ECHO + Practice Facilitation intervention.
  Charts included in this audit reflect an independent analytic sample of cancer survivors and do not necessarily represent the same individuals included in the baseline chart audit.
  Demographic characteristics were abstracted at this time point (Post) to describe the post-intervention sample.
  Analyses are descriptive and no inferential comparisons were conducted between baseline and post-intervention samples.
- Total: Total of all reporting groups
Arm/Group | Baseline (Pre-Intervention) Chart Audit | 24-Month Follow-Up (Post-Intervention) Chart Audit | Total
Number analyzed (Participants) | 138 | 129 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (mean and standard deviation) was abstracted from EHR charts included in the baseline sample (n=138). Values reflect age at the baseline pre-intervention period.
  years | 64.5 (7.7) | 63.0 (9.6) | 63.8 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was abstracted from EHR charts included in the baseline sample (n=138). Counts reflect the baseline pre-intervention period.
  Participants
    Female | 74 | 67 | 141
    Male | 64 | 62 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was abstracted from EHR charts included in the baseline sample (n=138) at the pre-intervention time point.
  Participants
    Hispanic or Latino | 3 | 3 | 6
    Not Hispanic or Latino | 121 | 125 | 246
    Unknown or Not Reported | 14 | 1 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was abstracted from EHR charts included in the baseline sample (n=138). Categories reflect OMB race classifications.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 130 | 96 | 226
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 2 | 30 | 32
Number of EHR charts analyzed at baseline [Number; unit: EHR charts] — "Participants" represent EHR charts selected for baseline analysis in a rural primary care survivorship intervention. No human participants were enrolled. Baseline characteristics reflect chart-level variables collected at the pre-intervention time point.
  EHR charts | 138 | 129 | 267

OUTCOME MEASURES:

1. Primary Outcome: Tumor Surveillance Completion (Pre-Intervention)
Description: This outcome reflects whether recommended tumor surveillance was completed and documented in the EHR. Tumor surveillance includes cancer-specific follow-up imaging consistent with evidence-based survivorship guidelines (e.g., NCCN, ASCO). Charts were coded as "Completed" if the recommended surveillance test was documented within the appropriate interval and "Not Completed" if documentation was absent, outdated, or incomplete. The outcome reports the proportion of EHR charts meeting tumor surveillance recommendations at baseline (pre-intervention) and again 24 months after the intervention.
Time Frame: Baseline (Pre-Intervention) Chart Audit
Population: Analysis population includes all EHR charts meeting inclusion criteria with complete documentation for the specified time point. Differences in sample size between baseline and post-intervention reflect routine variation in chart availability and completeness across clinics
Measure: Count of Participants; unit: Participants
Groups:
- KanSurvive ECHO + Practice Facilitation: This was a single-arm, delayed-start, clinic-level design. Primary care clinics were the unit of assignment and all clinics received the same KanSurvive ECHO + practice facilitation intervention. Pre- and post-intervention data represent chart abstractions, not longitudinal follow-up of the same individuals."
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 138
Participants | 126
Statistical Analysis 1: Comparison: KanSurvive ECHO + Practice Facilitation; Differences in cancer survivorship performance indicators and surveillance rates by tumor types before and after intervention were assessed using Fisher Exact tests; Test type: Other — Fisher Exact tests; p < 0.05, Chi-squared; Also used Fisher exact tests

2. Primary Outcome: Tumor Surveillance Completion (Post-Intervention)
Description: as for outcome 1
Time Frame: 24-Month Follow-Up (Post-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 129
Participants | 117

3. Primary Outcome: Distress Screening Completion (Pre-Intervention)
Description: This outcome reflects whether recommended Distress Screening was completed and documented in the EHR. Distress Screening was defined as documentation of using a standardized distress assessment tool consistent with survivorship best practices. Charts were coded as "Completed" when a distress screening result was documented during the chart abstraction interval. "Not Complete" indicated missing or incomplete documentation.
Time Frame: Baseline (Pre-intervention) Chart Review
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- KanSurvive ECHO + Practice Facilitation: This was a single-arm, delayed-start, clinic-level design. Primary care clinics were the unit of assignment and all clinics received the same KanSurvive ECHO + practice facilitation intervention. Pre- and post-intervention data represent chart abstractions, not longitudinal follow-up of the same individuals.
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 138
Participants | 116
Statistical Analysis 1: Comparison: KanSurvive ECHO + Practice Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Fisher exact tests; p < 0.05, Fisher Exact

4. Primary Outcome: Distress Screening Completion (Post-Intervention)
Description: as for outcome 3
Time Frame: 24-Month Follow-Up (Post-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 129
Participants | 116

5. Primary Outcome: Body Mass Index (BMI) Assessment Completion (Pre-Intervention)
Description: BMI assessment was defined as documentation of a height and weight measurement sufficient to calculate body mass index (BMI) in the electronic health record (EHR). Charts were coded as "Completed" when BMI or its components were documented within the recommended timeframe.
Time Frame: Baseline (Pre-intervention) Chart Review
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 138
Participants | 132
Statistical Analysis 1: Comparison: KanSurvive ECHO + Practice Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Fisher exact tests; p < 0.05, Fisher Exact

6. Primary Outcome: Body Mass Index (BMI) Assessment Completion (Post-Intervention)
Description: as for outcome 5
Time Frame: 24-Month Follow-Up (Post-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 129
Participants | 118

7. Primary Outcome: Tobacco Use Screening Completion (Pre-Intervention)
Description: Tobacco use screening was defined as documentation of current tobacco use status in the electronic health record (EHR). Charts were coded as "Completed" when a screening result was documented within the recommended timeframe.
Time Frame: Baseline (Pre-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 138
Participants | 115
Statistical Analysis 1: Comparison: KanSurvive ECHO + Practice Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Fisher exact test; p < 0.05, Fisher Exact

8. Primary Outcome: Tobacco Use Screening Completion (Post-Intervention)
Description: as for outcome 7
Time Frame: 24-Month Follow-Up (Post-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 129
Participants | 119

9. Primary Outcome: Cancer Diagnosis on Problem List (Pre-Intervention)
Description: This outcome reflects whether a cancer diagnosis was documented on the patient's EHR problem list, consistent with survivorship care documentation standards. Charts were coded as "Completed" when the cancer diagnosis appeared in the structured problem list.
Time Frame: Baseline (Pre-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 138
Participants | 129
Statistical Analysis 1: Comparison: KanSurvive ECHO + Practice Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Fisher exact test; p < 0.05, Fisher Exact

10. Primary Outcome: Cancer Diagnosis on Problem List (Post-Intervention)
Description: as for outcome 9
Time Frame: 24-Month Follow-Up (Post-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 129
Participants | 122

11. Primary Outcome: Family History of Cancer Documentation (Pre-Intervention)
Description: Family history of cancer documentation was defined as the presence of cancer-related family history information in the EHR. Charts were coded as "Completed" when documentation included a family history of cancer assessment entry.
Time Frame: Baseline (Pre-intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 138
Participants | 96
Statistical Analysis 1: Comparison: KanSurvive ECHO + Practice Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Fisher exact test; p < 0.05, Fisher Exact

12. Primary Outcome: Family History of Cancer Documentation (Post-Intervention)
Description: as for outcome 11
Time Frame: 24-Month Follow-Up (Post-Intervention) Chart Audit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KanSurvive ECHO + Practice Facilitation
Number analyzed (Participants) | 129
Participants | 115

ADVERSE EVENTS:
Time Frame: No adverse event monitoring was conducted because this was a retrospective EHR chart-review study with no enrolled patient participants.
Description: Because this study consisted solely of retrospective abstraction of electronic health record (EHR) data and did not involve prospective enrollment or exposure to an intervention, no adverse event assessments were performed. Adverse events were therefore not monitored or reported.
Groups:
- Baseline (Pre-Intervention) Chart Audit: Participants in this group represent independent EHR chart audit samples drawn from participating clinics.
- 24-Month Follow-Up (Post-Intervention) Chart Audit: Participants in this group represent independent EHR chart audit samples drawn from the same participating clinics.
  Cancer survivors charts included in the baseline (pre-intervention) chart audit are not necessarily the same cancer survivors included in the 24-month post-intervention chart audit.
  Therefore, the number of participants starting the post-intervention period is not expected to equal the number who completed the baseline period.
Arm/Group | Baseline (Pre-Intervention) Chart Audit | 24-Month Follow-Up (Post-Intervention) Chart Audit
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study relied on retrospective EHR abstraction in rural primary care practices, and documentation variability may not fully reflect all care delivered. Differences in baseline and post-intervention sample sizes reflect routine variation in chart availability and completeness. Data collection occurred during and following the COVID-19 pandemic, which affected project implementation, staffing and workflows.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04763824/Prot_SAP_000.pdf